CLINICAL TRIAL: NCT01654393
Title: Can Triage Nurse Initiated Radiographs in Accordance With the Ottawa Ankle Rule Shorten Emergency Department Length of Stay At a Tertiary Care Center?
Brief Title: Triage Nurse Initiated Radiographs According to OAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vancouver Coastal Health (Other Government)
Collaborators: University of British Columbia (Other)
Responsible Party: Principal Investigator, Dr. Lyne Filiatrault, Emergency Physician, Vancouver Coastal Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: H12-01352
Record Dates: First submitted 2012-07-27; First posted 2012-07-31 (Estimated); Last update posted 2012-09-12 (Estimated); Status verified 2012-09

CONDITIONS: Ankle Fracture
Keywords: Triage nurse; Ottawa ankle rules
MeSH Terms: conditions — Ankle Fractures

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- OAR group (Experimental): Patients with ankle injuries who are assessed by OAR trained triage nurses applying the OAR.
  Interventions: Other: Triage nurses applying the OAR
- Control for OAR Triage Nurses (No Intervention): Patients with ankle injuries that are seen by OAR triage nurses but not assessed in accordance with the OAR.

INTERVENTIONS:
Other: Triage nurses applying the OAR — Triage nurses applying the OAR during assessment and ordering foot/ankle x-rays as necessary.
  Arms: OAR group

SUMMARY:
The purpose of the study is to help doctors in emergency departments know whether triage nurse initiated radiographs, in accordance to the Ottawa ankle rule, before emergency physician assessment will shorten emergency patients' visit. The investigators will examine the number of missed fractures between the two groups, the emergency physicians' willingness to apply OAR and triage nurses' satisfaction.

DETAILED DESCRIPTION:
Overcrowding in the emergency department (ED) has been an ongoing issue for many hospitals in North America. Numerous strategies have been implemented and explored in hopes of reducing wait times and length of stay. The Ottawa ankle rules are one such strategy developed and proven to reduce cost and wait time without patient dissatisfaction and missed fractures. As a result, they have gained widespread acceptance from emergency physicians around the world.

Since the implementation of the Ottawa ankle rules (OAR), numerous studies have examined nurses' application and interpretation of these rules. It has been shown that nurses' application of the rule yield similar sensitivity and negative predictability for diagnosis of fractures as physicians. It is believed that emergency nurses can make accurate assessment in the determination of the patients who require radiographs. What is unclear, however, is whether or not triage nurse initiated radiographs shortens patients' length of stay in the emergency department, a factor inversely correlated to patient satisfaction. Only a couple of studies have looked at this issue in the context of the Ottawa ankle rules. One is a retrospective study conducted at an A&E department in a small city while the other, although randomized prospectively, was carried out in an urgent care center rather than in a busy academic tertiary care hospital.

Our primary objective for this study is to investigate the median length of stay of patients presenting to a tertiary care academic center with blunt ankle injuries and assess whether triage nurse initiated radiographs in accordance to the Ottawa ankle rules would shorten their stay versus current standard of care. Presently, the emergency physician orders the x-ray at the time of patient encounter.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 19 presenting with an isolated blunt ankle injury

Exclusion Criteria:

* Injury >10 days
* Isolated skin injury
* Referred patient with outside x-ray
* Obvious fracture or deformity
* Polytrauma
* Pregnancy
* Diminished sensation due to neurological deficit
* Uncooperative, intoxicated or patients with altered mental status
* Patients returning for reassessment of same injury
* Injury due to or suspicious for domestic violence

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-01 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
Median length of stay (LOS) of patients presenting to a tertiary care academic center with blunt ankle injuries | 6 months
  Median LOS will be measured and compared among patients with ankle injuries that were assessed by OAR trained triage nurses who applied the OAR and ordered X-rays if necessary vs those patients who were triaged as per usual practice, with no OAR application.

SECONDARY OUTCOMES:
Fracture missed by Triage Nurse: | Estimated at 6 months.
  Assess if fractures were missed by triage nurse via + X-rays ordered by EP or via follow-up questionnaire 2 weeks later to determine if other investigations were performed after the pt's visit to the ED
Triage nurses' satisfaction | estimated at 6 months
  Assess triage nurse' feedback regarding comfortability in applying the OAR, training, and whether the OAR has increased workload.
Percent agreement regarding necessity for X-ray between emergency nurse and physician | estimated at 6 months
Emergency physician's compliance with OAR | estimated at 6 months
  Determine if emergency physicians are applying OAR during this study period
Patient satisfaction with triage nurse initiated imaging | Estimated at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Lyne Filiatrault, MD, FRCPC, Principal Investigator — Vancouver Coastal Health Authorities; Wailliam W Lee, MD, Principal Investigator — Vancouver Costal Health Authorities; Ryiad Abu-Laban, MD, MHSc, FRCPC, Principal Investigator — Vancouver Costal Health Authorities
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada